CLINICAL TRIAL: NCT03769675
Title: Quantitative Assessment of Painful Diabetic Peripheral Neuropathy After High Frequency Spinal Cord Stimulation: (QUANT) HF10 Study
Brief Title: Quantitative Assessment of Painful Diabetic Peripheral Neuropathy After High Frequency Spinal Cord Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Narayan R. Kissoon, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-004317
Record Dates: First submitted 2018-11-20; First posted 2018-12-07 (Actual); Results first posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Painful Diabetic Neuropathy
Keywords: spinal cord stimulation; type 2 diabetes
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Spinal Cord Stimulator Implant (Experimental): Spinal Cord Stimulator implant
  Interventions: Device: High Frequency Spinal Cord Stimulator

INTERVENTIONS:
Device: High Frequency Spinal Cord Stimulator — The SCS implant will follow standard clinical practice for these FDA approved indications. Two percutaneous leads will be placed in the posterior spinal epidural space under radiographic guidance and attached to either an external stimulator (trial phase) or a subcutaneously implanted impulse generator (IPG). Intraoperative impedance testing will be performed to ensure electrical integrity. Patients with HF10 SCS will receive 30 µs pulses delivered at 10,000 Hz with amplitude adjusted to optimal analgesic response. Programming will occur postoperatively and as needed based on patient feedback in standard clinic visits. .

SUMMARY:
Will participants with painful lower extremity diabetic peripheral neuropathy (DPN) that are treated with high frequency spinal cord stimulation (HF10 SCS) have improvements in lower extremity peripheral nerve function?

DETAILED DESCRIPTION:
This research study is being conducted to find out if spinal cord stimulation (SCS) can improve nerve function. SCS is FDA approved for the treatment of intractable neuropathic (nerve) pain related to diabetic peripheral neuropathy. With SCS a wire is placed in the epidural space and the spinal cord is stimulated to interrupt the pain signal coming from the legs. The spinal cord stimulator is a device similar to a pacemaker (which helps treat abnormal rhythms of the heart). Recent studies have suggested that SCS with high frequencies can improve nerve function for subjects with painful peripheral neuropathy therefore, the investigators are looking to measure changes in nerve function after SCS for treatment of painful diabetic peripheral neuropathy.

The purpose of this research is to gather information on the effect of high frequency spinal cord stimulation (HF10) on nerve function with a spinal cord stimulator.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Refractory predominantly lower extremity neuropathic pain for > 1 year
* Presence of length dependent peripheral neuropathy on sudomotor testing
* Completed spinal cord stimulation trial with 40% or greater pain reduction from baseline
* Failed medication trials or contraindication to gabapentin medications (gabapentin, pregabalin) and/or serotonin/norepinephrine reuptake inhibitors (tricyclic antidepressant (TCA) or duloxetine or venlafaxine)
* Average pain score on a visual analog scale (VAS) of ≥ 5 (with 0 representing no pain and 10 the worst pain imaginable)
* Appropriate surgical candidate for spinal cord stimulator

Exclusion Criteria:

* Severe Autonomic Neuropathy as measured by the composite autonomic scoring scale (10 point scale) with a score ≥ 7
* History of sympathectomy
* Uncontrolled arterial hypertension (Systolic Blood Pressure >160)
* Baseline Foot TcPO2 < 10 mmHg to exclude patients with severe peripheral arterial disease
* Hemoglobin A1c > 8%
* Stable opioid regimen with oral morphine equivalent ≥ 100 mg/day
* Alternative principle cause for peripheral neuropathy or lower extremity neuropathic pain
* Disruptive psychiatric disorder (screened for during preoperative psychiatric evaluation)
* Pending litigations
* Women of child bearing potential unwilling to use contraception or found to be pregnant as part of perioperative screening
* Patients unable to hold medications that would impact autonomic testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Narayan R Kissoon, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Kissoon NR, LeMahieu AM, Stoltenberg AD, Bendel MA, Lamer TJ, Watson JC, Sletten DM, Singer W. Quantitative assessment of painful diabetic peripheral neuropathy after high-frequency spinal cord stimulation: a pilot study. Pain Med. 2023 Oct 13;24(Suppl 2):S41-S47. doi: 10.1093/pm/pnad087. PMID 37833046
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Spinal Cord Stimulator Implant (SCS): Spinal Cord Stimulator implant
  High Frequency Spinal Cord Stimulator: The SCS implant followed standard clinical practice for FDA approved indications: Two percutaneous leads were placed in the posterior spinal epidural space under radiographic guidance and attached to either an external stimulator or a subcutaneously implanted impulse generator (IPG). Intraoperative impedance testing was performed to ensure electrical integrity. Patients with HF10 SCS received 30 µs pulses delivered at 10,000 Hz with amplitude adjusted to optimal analgesic response. Programming occurred postoperatively and as needed based on patient feedback in standard clinic visits.
Period: Overall Study
Arm/Group | Spinal Cord Stimulator Implant (SCS)
Started | 10
Completed | 9
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Spinal Cord Stimulator Implant (SCS)
Number analyzed (Participants) | 10
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55.0 [48.0 to 61.0]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
  F-Transgender | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Pain Assessment
Description: Pain measurement using a Visual Analog Pain Scale by placing an X in the box to indicate the severity of pain from no pain to intolerable pain. The X in the box translates to a score of zero for no pain and increases by an additional 0.5 up to a high score of 10 which would be intolerable pain.
Time Frame: Baseline, 12 months
Population: Data was not collected or analyzed at 12 months for the one subject who did not complete the study.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Spinal Cord Stimulator Implant (SCS)
Number analyzed (Participants) | 10
score on a scale
  baseline | 6.5 [5.0 to 8.0]
  12 months: number analyzed (Participants) | 9
  12 months | 1.0 [1.0 to 3.0]

2. Primary Outcome: Neuropathy Symptoms and Change (NSC) Score
Description: Validated questionnaire that evaluates change in neuropathy symptoms, including symptoms of weakness, sensory symptoms, and autonomic symptoms. Answers to questionnaire are yes/no and if yes, then degree of severity is evaluated with a plus one(slight), plus two (moderate) and plus three (severe). Questionnaire screens the presence and severity of diabetic peripheral neuropathy. Change in severity of symptoms are compared over time. Total scores range from 0 - 114, lower scores reflect no neuropathy symptoms, higher scores reflect more neuropathy symptoms.
Time Frame: baseline, 12 months
Population: Data was not collected or analyzed at 12 months for the one subject who did not complete the study.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Spinal Cord Stimulator Implant (SCS)
Number analyzed (Participants) | 10
score on a scale
  baseline | 21.5 [16.0 to 28.0]
  12 months: number analyzed (Participants) | 9
  12 months | 9.0 [6.0 to 12.0]

3. Primary Outcome: Oswestry Disability Index
Description: Questionnaire examines perceived level of disability in 10 everyday activities of daily living including pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life and traveling. The 6 statements are scored from 0 to 5 scale, zero meaning no disability. The final score ranges from 0-100 with a score of 0-20 equals minimal disability, 21-40 equals moderate disability, 41-60 equals severe disability, 61-80 equals crippled and 81-100 equals bed-bound.
Time Frame: Baseline, 12 months
Population: Data was not collected or analyzed at 12 months for the one subject who did not complete the study.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Spinal Cord Stimulator Implant (SCS)
Number analyzed (Participants) | 10
score on a scale
  baseline | 37.0 [28.0 to 56.0]
  12 months: number analyzed (Participants) | 9
  12 months | 18.0 [12.0 to 40.0]

4. Primary Outcome: Neuropathy Impairment Score (NIS)
Description: Subject's scores neuropathic deficits using a scale of 0-4 (zero=normal, 4=paralysis) to measure muscle weakness. The NIS score is a measure of neurologic impairment. The NIS Score has a range of 0 to 244. Lower scores indicate higher function, higher scores indicate lower function.
Time Frame: Baseline, 12 months
Population: Data was not collected or analyzed at 12 months for the one subject who did not complete the study.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Spinal Cord Stimulator Implant (SCS)
Number analyzed (Participants) | 10
score on a scale
  baseline | 15.0 [12.0 to 24.0]
  12 months: number analyzed (Participants) | 9
  12 months | 13.0 [6.0 to 16.0]

5. Primary Outcome: Lower Limb Function Test
Description: Test for lower limb function in which the subject will need to walk on toes, walk on heels, and arise from kneeled position, each test is marked as not applicable, normal or abnormal. The examination assesses each component for the left and right side separately. If the test is normal, it is given a score of 0, and if it is abnormal, a score of 1. Not applicable scores a zero. Total scores range 0-6. Therefore, the maximum score of 6 indicates abnormality in all 3 components bilaterally and a minimum score of 0 indicates a normal result for all 3 components bilaterally.
Time Frame: Baseline, 12 months
Population: Data was not collected or analyzed at 12 months for the one subject who did not complete the study.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Spinal Cord Stimulator Implant (SCS)
Number analyzed (Participants) | 10
score on a scale
  Baseline | 1 [0 to 2]
  12 months: number analyzed (Participants) | 9
  12 months | 0 [0 to 0.5]

6. Primary Outcome: Modified Leads Assessment of Neuropathic Symptoms and Signs
Description: Questionnaire to identify and analyze pain by answering yes/no which translates to scores from 0-24. A score of 12 or more suggests pain of predominantly neuropathic origin.
Time Frame: baseline, 12 months
Population: Data was not collected or analyzed at 12 months for the one subject who did not complete the study.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Spinal Cord Stimulator Implant (SCS)
Number analyzed (Participants) | 10
score on a scale
  baseline | 19.0 [16.0 to 24.0]
  12 months: number analyzed (Participants) | 9
  12 months | 17.0 [11.0 to 22.0]

7. Primary Outcome: Positive Pain
Description: Numeric Rating Scale used to assess pain from a scale of 0 (no pain) to 10 (worst possible pain)
Time Frame: baseline, 12 months
Population: Data was not collected or analyzed at 12 months for the one subject who did not complete the study.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Spinal Cord Stimulator Implant (SCS)
Number analyzed (Participants) | 10
score on a scale
  baseline | 9.0 [8.0 to 10.0]
  12 months: number analyzed (Participants) | 9
  12 months | 3.0 [2.0 to 4.0]

8. Secondary Outcome: Patient Health Questionnaire
Description: Screens for the presence and severity of depression with 9 questions in a scale of 0-3. Zero=not at all, 1=several days, 2=more than half the days, 3=nearly every day. Total score range 0 - 27. A total score of 0-4=minimal depression, 5-9=mild depression, 10-14=moderate depression, 15-19=moderately severe depression, 20-27=severe depression
Time Frame: Baseline, 12 months
Population: Data was not collected or analyzed at 12 months for the one subject who did not complete the study.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Spinal Cord Stimulator Implant (SCS)
Number analyzed (Participants) | 10
score on a scale
  baseline | 4.0 [3.0 to 12.0]
  12 months: number analyzed (Participants) | 9
  12 months | 2.0 [2.0 to 6.0]

9. Secondary Outcome: Height
Description: Subjects calculated height in centimeters.
Time Frame: Baseline, 12 months
Population: Data was not collected or analyzed at 12 months for the one subject who did not complete the study.
Measure: Median (Inter-Quartile Range); unit: cm
Arm/Group | Spinal Cord Stimulator Implant (SCS)
Number analyzed (Participants) | 10
cm
  baseline | 173 [160 to 185]
  12 months: number analyzed (Participants) | 9
  12 months | 175 [159 to 186]

10. Secondary Outcome: Weight
Description: Subjects calculated weight in kilograms
Time Frame: Baseline, 12 months
Population: Data was not collected or analyzed at 12 months for the one subject who did not complete the study.
Measure: Median (Inter-Quartile Range); unit: kg
Arm/Group | Spinal Cord Stimulator Implant (SCS)
Number analyzed (Participants) | 10
kg
  baseline | 97.0 [85.3 to 107.0]
  12 months: number analyzed (Participants) | 9
  12 months | 97.2 [92.9 to 123.0]

11. Secondary Outcome: Body Mass Index (BMI)
Description: Subject's BMI calculated as weight in kilograms divided by height in meters squared. Uses measurements of height and weight obtained during study (with appropriate metric conversions)
Time Frame: Baseline, 12 months
Population: Data was not collected or analyzed at 12 months for the one subject who did not complete the study.
Measure: Median (Inter-Quartile Range); unit: kg/m^2
Arm/Group | Spinal Cord Stimulator Implant (SCS)
Number analyzed (Participants) | 10
kg/m^2
  baseline | 34.3 [31.2 to 36.1]
  12 weeks: number analyzed (Participants) | 9
  12 weeks | 34.5 [31.2 to 37.3]

12. Secondary Outcome: Hemoglobin A1c
Description: Hemoglobin is a protein within red blood cells. As glucose enters the bloodstream, it binds to hemoglobin, or glycates. The more glucose that enters the bloodstream, the higher the amount of glycated hemoglobin. An A1C level below 5.7 percent is considered normal. Reported as percentage of glycated hemoglobin
Time Frame: Baseline, 12 months
Population: Data was not collected or analyzed at 12 months for the one subject who did not complete the study.
Measure: Median (Inter-Quartile Range); unit: percentage of glycated hemoglobin
Arm/Group | Spinal Cord Stimulator Implant (SCS)
Number analyzed (Participants) | 10
percentage of glycated hemoglobin
  baseline | 7.3 [6.1 to 7.7]
  12 weeks: number analyzed (Participants) | 9
  12 weeks | 7.85 [6.2 to 8.6]

13. Secondary Outcome: Forearm Sweat Volume Quantitative Axon Reflex Sweat Test (Q-SWEAT)
Description: Test that measures the rate and volume of sweat to determine the severity and pattern of autonomic disorders. As measured by µL/cm²
Time Frame: baseline, 12 months
Population: Data was not collected or analyzed at 12 months for the one subject who did not complete the study.
Measure: Median (Inter-Quartile Range); unit: µL/cm²
Arm/Group | Spinal Cord Stimulator Implant (SCS)
Number analyzed (Participants) | 10
µL/cm²
  baseline | 1.3 [0.3 to 1.9]
  12 months: number analyzed (Participants) | 9
  12 months | 0.3 [0.2 to 1.6]

14. Secondary Outcome: Proximal Leg Laser Doppler Flowmetry (LDF)
Description: Laser Doppler velocimetry is used in hemodynamics research as a technique to partially quantify blood flow in human tissues such as skin. Within the clinical environment, the technology is often referred to as laser Doppler flowmetry (LDF). As measured in perfusion units (p.u.)
Time Frame: Baseline, 12 months
Population: Data was not collected or analyzed at 12 months for the one subject who did not complete the study.
Measure: Median (Inter-Quartile Range); unit: perfusion units (p.u.)
Arm/Group | Spinal Cord Stimulator Implant (SCS)
Number analyzed (Participants) | 10
perfusion units (p.u.)
  baseline | 22.2 [14.7 to 28.3]
  12 months: number analyzed (Participants) | 9
  12 months | 29.0 [18.8 to 29.8]

15. Secondary Outcome: Extensor Digitorum Brevis Muscle Nerve Conduction
Description: A nerve conduction study (NCS) is a medical diagnostic test commonly used to evaluate the function, especially the ability of electrical conduction, of the motor and sensory nerves of the human body. As measured by amplitude (AMP) milliamp (mA)
Time Frame: Baseline, 12 months
Population: Data was not collected or analyzed at 12 months for the one subject who did not complete the study.
Measure: Median (Inter-Quartile Range); unit: AMP (mA)
Arm/Group | Spinal Cord Stimulator Implant (SCS)
Number analyzed (Participants) | 10
AMP (mA)
  baseline | 3.1 [0.6 to 5.1]
  12 months: number analyzed (Participants) | 9
  12 months | 1.0 [0.5 to 5.0]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to end of study, approximately 12 months
Arm/Group | Spinal Cord Stimulator Implant (SCS)
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-27): https://cdn.clinicaltrials.gov/large-docs/75/NCT03769675/Prot_SAP_000.pdf